CLINICAL TRIAL: NCT04994873
Title: Skills to Enhance Positivity in Adolescents at Risk for Suicide
Brief Title: Skills to Enhance Positivity in Suicidal Youth
Acronym: STEP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Anthony Spirito, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1023
Record Dates: First submitted 2021-07-25; First posted 2021-08-06 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-06

CONDITIONS: Suicide, Attempted
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: 2 condition randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: The baseline assessment will occur prior to randomization and follow-up assessors will be blind to participant condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEP: Positivity skill enhancement (Experimental): This intervention includes the Enhanced TAU described below plus it entails 4 in-person sessions delivered during an inpatient psychiatric admission, followed by mood monitoring and skills messages delivered post-discharge via app, to promote the practice of increasing attention to positive affect and experiences as a means of reducing risk for suicidal behavior.
  Interventions: Behavioral: STEP
- Enhanced TAU (Active Comparator): his comparison intervention involves regular programming of the inpatient psychiatric unit, followed by safety plan and resources loaded onto an app that the participant has access to post-discharge.
  Interventions: Behavioral: Enhanced TAU

INTERVENTIONS:
Behavioral: STEP — Behavioral intervention to increase positive affect
  Arms: STEP: Positivity skill enhancement
Behavioral: Enhanced TAU — Standard care plus a phone app with a personalized safety plan
  Arms: Enhanced TAU

SUMMARY:
This is a Hybrid Type I Effectiveness-Implementation design. Specifically, this study proposes to test the effectiveness of STEP in reducing suicidal events and ideation in 216 adolescents, admitted to inpatient psychiatric care due to suicide risk. Participants will be randomized to either STEP or ETAU. STEP involves 4 in-person sessions (3 individual, 1 family) focused on psychoeducation regarding positive and negative affect, mindfulness meditation, gratitude, and savoring. Mood monitoring prompts and skill reminders will be sent daily for the first month post-discharge and three times a week for the following two months. The ETAU condition will receive reminders to log into a safety resource app, matched in frequency to the STEP group. Effectiveness aspects of the design include using clinical staff as interventionists and having very few exclusion criteria.

DETAILED DESCRIPTION:
216 participants and their families (across two sites) will be randomized to either STEP or ETAU (as described in the research strategy). Aims and hypotheses are below:

Aim 1: Examine the effectiveness of STEP in reducing suicidal events (attempt or emergency intervention to intercede attempt), active SI (with intent or plan), and depression at 6-month f/u (primary) and suicidal events at 12-month follow-up (f/u). H1: It is hypothesized that those randomized to STEP, compared to ETAU, will have lower rates of suicide events (H1A), active SI (H1B), and depression (H1C) over the 6-month follow-up period; H1D: It is hypothesized that those randomized to STEP, compared to ETAU, will have lower rates of suicidal events at the 12-month, long term f/u.

Aim 2: Examine engagement of the hypothesized mechanisms at the 3- and 6-month f/u. It is hypothesized that those randomized to STEP, compared to ETAU, will have: H2A: higher attention to positive affect, assessed by implicit tasks; H2B: higher gratitude and satisfaction with life, assessed by self-report; H2C: lower negative affect, assessed by implicit tasks and self-report.

Aim 3: Examine whether hypothesized mechanisms mediate reduction of suicidal events and ideation. H3: Changes in attention to positive affect, gratitude, satisfaction with life, and negative affect at 3-month f/u will be related to improvements in suicidal ideation and suicidal events at the 6-month f/u.

Secondary Aim Examine elements supporting external validity. Acceptability, appropriateness, and feasibility of STEP to patients, parents, clinicians, and administrators will be assessed by: 1) a survey consisting of brief, standardized measures of these items, and 2) qualitative interviews to further explore these perceptions. These findings will be used to: 1) modify STEP to address potential barriers, and 2) develop implementation strategies designed to overcome these challenges, for testing in a future Hybrid Type III effectiveness-implementation trial.

ELIGIBILITY:
Inclusion Criteria: Patients

* Ages 12- 60 years
* hospitalized on an inpatient psychiatric unit due to suicide risk
* past month suicide attempts or suicidal ideation
* proficient in English (parent either English or Spanish
* access to a smart phone.

Inclusion Criteria: Stakeholders

Ages 22 - 60 years

* work with adolescents hospitalized on an inpatient psychiatric unit due to suicide risk
* proficient in English or Spanish

Exclusion Criteria:

* active psychotic disorder
* significant cognitive impairment or deficits
* ward of the State
* discharge to residential facility.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Suicidal events | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Composite variable of either a suicide attempt or emergency intervention to intercede when suicidal behavior may be imminent; Will be obtained from clinical interviews (C-SSRS; CASA) with the participant and parent(s).
Suicidal ideation | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Suicide Ideation (SI) will be operationalized as proportion of participants with active SI as assessed by the Columbia Suicide Severity Rating Scale interview: 5 items on suicidal ideation rated yes or no
Proportion of Weeks with Suicidal ideation | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  The proportion of weeks during follow-up with active suicidal ideation as assessed by the Adolescent version of the Longitudinal Interview for Follow-Up Events (A-LIFE) scale (interview based assessment), with the participant.
Depression | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Depressive symptom severity will be assessed using the Beck Depression Inventory II (BDI-II). The BDI-II will be administered to the adolescent participant and their parent (reporting on the adolescent participant) with scores ranging from 0 to 63 with higher scores reflecting greater depression.

SECONDARY OUTCOMES:
Attention to positive affect | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Using eye tracking we will measure fixation and overall gaze duration during a dot probe task using emotional and neutral words to determine whether there is a change in attention to positive affect (participant only).
Implicit positive and negative affect | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Implicit positive affect will be assessed using the Implicit Positive and Negative Affect Test (IPANAT), which is an indirect assessment of automatic activation of affective representations that utilizes artificial words paired with positive and negative words (participant only).
Explicit positive and negative affect | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Explicit positive affect will be assessed using the Modified Differential Emotions Scale (mDES) which is a 20 item short term self-report of positive and negative emotions administered to the participant only. There are 10 items in the positive affect and 10 items in the negative affect subscales with scores ranging from 0 to 30 for each subscale with higher scores reflecting higher affect.
Gratitude | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  Gratitude will be assessed with the 6 item Gratitude Scale, administered to the participant only. Scores range from 6 to 42 with higher scores indicating greater gratitude.
Satisfaction with life scale | baseline; change from baseline at 3 months, 6 months, and 12 months follow-up
  5 self-report questions about participant satisfaction with life with scores ranging from 7 to 35 with higher scores indicating higher satisfaction with life.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Children's Hospital, Boston, Massachusetts
  - Butler Hospital, Providence, Rhode Island
  - Bradley Hospital, Riverside, Rhode Island

IPD SHARING:
Plan to Share IPD: Yes
We will release demographics, primary and secondary data thru the NDA
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Final data set available within one year of completion
Access Criteria: University-based researchers

REFERENCES:
- [Derived] Yen S, Suazo N, Doerr J, Macrynikola N, Villarreal LS, Sodano S, O'Brien KHM, Wolff JC, Breault C, Gibb BE, Elwy R, Kahler CW, Ranney M, Jones R, Spirito A. Skills to Enhance Positivity in adolescents at risk for suicide: Protocol for a randomized controlled trial. PLoS One. 2023 Oct 20;18(10):e0287285. doi: 10.1371/journal.pone.0287285. eCollection 2023. PMID 37862324